CLINICAL TRIAL: NCT02756611
Title: Open-Label, Single Arm, Phase 3b, Multi-Center Study Evaluating the Efficacy of Venetoclax (ABT 199) in Relapsed/Refractory Subjects With Chronic Lymphocytic Leukemia (CLL)
Brief Title: A Study to Evaluate the Efficacy of Venetoclax Monotherapy in Relapsed/Refractory Participants With Chronic Lymphocytic Leukemia (CLL)
Acronym: VENICE I
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M15-550; 2015-003667-11 (EudraCT Number)
Expanded Access: NCT03123029 (Available)
Record Dates: First submitted 2016-04-26; First posted 2016-04-29 (Estimated); Results first posted 2020-05-04 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-04

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: Oncology; Chronic Lymphocytic Leukemia; 17p Deletion; TP53 Mutation; Relapsed; Refractory; B-Cell receptor inhibitor
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Neoplasms; Chromosome 17 deletion; Recurrence | interventions — venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Venetoclax (Experimental): Venetoclax will be administered orally once daily (QD) beginning with a dose-titration phase. The initial venetoclax dose is 20 mg QD. After 1 week of treatment at 20 mg QD, the dose will be escalated to 50 mg QD followed by subsequent increases, each after 1 week, to 100 mg QD, 200 mg QD and the maximum dose of 400 mg QD. Participants may continue to receive venetoclax for up to 2 years provided they continue to tolerate the drug, have no evidence of disease progression (based on investigator's assessment), do not have unacceptable toxicity, and do not meet any of the criteria for discontinuation.
  In countries where venetoclax is not commercially available, participants who continue to derive benefit after 2 years of treatment may be able to extend their treatment for up to 2 additional years, plus one additional year until the venetoclax extension study was open, determined on a case by case basis.
  Interventions: Drug: Venetoclax

INTERVENTIONS:
Drug: Venetoclax — Tablets for oral administration
  Other Names: ABT-199; VENCLEXTA®

SUMMARY:
The purpose of this study is to evaluate the efficacy of venetoclax monotherapy in participants with relapsed/refractory CLL with or without the 17p deletion or TP53 mutation, including those who have received prior treatment with a B-cell receptor inhibitor.

DETAILED DESCRIPTION:
Following the Screening period, all eligible participants initiate venetoclax on a once daily (QD) dosing schedule. To mitigate the risk for tumor lysis syndrome (TLS), dosing will start with a 5-week dose titration phase.

Participants may receive venetoclax for up to 2 years provided they continue to tolerate the drug, have no evidence of disease progression (based on investigator assessment), do not have unacceptable toxicity and do not meet any of the criteria for subject discontinuation. In countries where venetoclax is not commercially available, participants who continued to derive benefit after 2 years of treatment may extend their treatment for up to 2 additional years in an extended access phase. Participants in the extended access phase of this study who continue to derive benefit from venetoclax after the 2-year extension and are transferring to the venetoclax extension study, Study M19-388 (NCT03844048), may remain in Extended Access for up to 1 additional year or until the extension study is approved and initiated at the site, whichever is sooner.

ELIGIBILITY:
Inclusion Criteria:

* Participant has Eastern Cooperative Oncology Group (ECOG) performance score of less than or equal to 2
* Participant has relapsed/refractory disease (received at least 1 prior therapy)
* Participant has diagnosis of CLL that meets published 2008 Modified International Workshop for Chronic Lymphocytic Leukemia National Cancer Institute Working Group (IWCLL NCI-WG) Guidelines and:

  * has an indication for treatment according to the 2008 Modified IWCLL NCI-WG criteria
  * has clinically measurable disease (lymphocytosis greater than 5 × 10^9/L and/or palpable and measurable nodes by physical exam and/or organomegaly assessed by physical exam)
* In addition, participants:

  * with or without 17p deletion or TP53 mutation, assessed by a local laboratory in bone marrow or peripheral blood are eligible
  * may have been previously treated with a prior B-cell receptor inhibitor
* Participant must have adequate bone marrow function, coagulation profile, renal, and hepatic function, per laboratory at Screening

Exclusion Criteria:

* Participant has developed Richter's transformation or Prolymphocytic leukemia
* Participant has previously received venetoclax
* History of active malignancies other than CLL within the past 2 years prior to first dose of venetoclax, with the exception of:

  * adequately treated in situ carcinoma of the cervix uteri
  * adequately treated basal cell carcinoma or localized squamous cell carcinoma of the skin
  * previous malignancy confined and surgically resected (or treated with other modalities) with curative intent
* Participant has active and uncontrolled autoimmune cytopenias (for 2 weeks prior to Screening), including autoimmune hemolytic anemia and idiopathic thrombocytopenic purpura despite low dose corticosteroids
* Participant has undergone an allogeneic stem cell transplant
* Treatment with any of the following within five half-lives or 14 days (if half-life unknown) as applicable prior to the first dose of venetoclax, or clinically significant adverse effect(s)/toxicity(s) of the previous therapy have not resolved to < National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v4.03 Grade 2:

  * Any anti-cancer therapy including chemotherapy, or radiotherapy;
  * Investigational therapy, including targeted small molecule agents
* Participant is human immunodeficiency virus (HIV) positive
* Participant has known allergy to both xanthine oxidase inhibitors and rasburicase

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Actual)
Dates: Start 2016-06-22 (Actual); Primary Completion 2019-04-10 (Actual); Study Completion 2022-03-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (67):
- United States (6):
  - Norton Cancer Institute /ID# 149788, Louisville, Kentucky
  - St. Agnes Cancer Center /ID# 149782, Baltimore, Maryland
  - Hackensack Univ Med Ctr /ID# 151574, Hackensack, New Jersey
  - Utah Cancer Specialists /ID# 151604, Salt Lake City, Utah
  - Cancer Care Northwest /ID# 151605, Spokane, Washington
  - West Virginia Univ School Med /ID# 151602, Morgantown, West Virginia
- Austria (3):
  - LKH-Univ. Klinikum Graz /ID# 147547, Graz
  - LKH Salzburg and Paracelsus /ID# 147549, Salzburg
  - Hanusch Krankenhaus der WGKK /ID# 147548, Vienna
- Belgium (2):
  - Cliniques Universitaires Saint Luc /ID# 147388, Woluwe-Saint-Lambert, Brussels Capital
  - UZ Leuven /ID# 147387, Leuven
- Canada (5):
  - BC Cancer Agency /ID# 153091, Vancouver, British Columbia
  - Qe Ii Hsc /Id# 147460, Halifax, Nova Scotia
  - Juravinski Cancer Clinic /ID# 149152, Hamilton, Ontario
  - Sunnybrook Health Sciences Ctr /ID# 147462, Toronto, Ontario
  - CHU de Quebec-Universite Laval /ID# 150299, Québec, Quebec
- Denmark (2):
  - Herlev Hospital /ID# 150183, Herlev, Capital Region
  - Aarhus University Hospital /ID# 147409, Aarhus N, Central Jutland
- Turku University Hospital /ID# 147551, Turku, Finland
- France (5):
  - CHU Dupuytren /ID# 147552, Limoges, Franche-Comte
  - CHU de la miletrie /ID# 147484, Poitiers, Poitou-Charentes
  - Institut Bergonie /ID# 147482, Bordeaux
  - CHRU de Brest - Hopital Morvan /ID# 147485, Brest
  - clinique Sainte Anne /ID# 147556, Strasbourg
- Germany (5):
  - Onkologische Schwerpunktpraxis /ID# 147516, Berlin
  - Cent fuer Haematologie und Onk /ID# 147511, Frankfurt
  - OncoResearch Lerchenfeld GmbH /ID# 164044, Hamburg
  - Mannheimer Onkologiepraxis /ID# 147512, Mannheim
  - Staedt. Klinikum Schwabing /ID# 147510, Munich
- Greece (2):
  - General Hospital of Athens Laiko /ID# 147517, Athens, Attica
  - G. Papanikolaou Hospital /ID# 147518, Thessaloniki
- Ireland (2):
  - St. James's Hospital /ID# 147519, Dublin, Dublin
  - Beaumont Hospital /ID# 147522, Dublin
- Israel (3):
  - Tel Aviv Sourasky Medical Ctr /ID# 151624, Tel Aviv, Tel Aviv
  - Galilee Medical Center /ID# 159971, Nahariya
  - Sheba Medical Center /ID# 147509, Ramat Gan
- Italy (5):
  - A.O.U. Policlinico S.Orsola-Malpighi /ID# 147505, Bologna, Emilia-Romagna
  - AP Romano Umberto I /ID# 147500, Rome, Lazio
  - ASST Grande Ospedale Metropolitano Niguarda /ID# 147503, Milan, Lombardy
  - Ospedale San Raffaele IRCCS /ID# 147504, Milan
  - AO Maggiore della Carita /ID# 147499, Novara
- Netherlands (2):
  - Academisch Medisch Centrum /ID# 147494, Amsterdam, North Holland
  - Albert Schweitzer Ziekenhuis /ID# 147495, Dordrecht, South Holland
- Norway (2):
  - Haukeland University Hospital /ID# 147382, Bergen, Hordaland
  - Rikshospitalet OUS HF /ID# 201812, Oslo
- Portugal (2):
  - IPO Lisboa FG, EPE /ID# 147385, Lisbon
  - IPO Porto FG, EPE /ID# 147389, Porto
- Puerto Rico Hematology Oncolog /ID# 150003, San Juan, Puerto Rico
- Spain (5):
  - Hospital Santa Creu i Sant Pau /ID# 151230, Barcelona
  - Fundacion Jimenez Diaz /ID# 151231, Madrid
  - Hosp Univ Puerta de Hierro /ID# 147391, Majadahonda
  - Hospital Clinico Univ de Salamanca /ID# 147392, Salamanca
  - Hosp Clin Univ de Valencia /ID# 147396, Valencia
- Sweden (2):
  - Skanes Universitetssjukhus Lund /ID# 147439, Lund, Skåne County
  - Akademiska Sjukhuset /ID# 150184, Uppsala, Uppsala County
- Switzerland (3):
  - Hopitaux Universitaires de Geneve /ID# 147930, Geneva, Canton of Geneva
  - University Hospital Zurich /ID# 157910, Zurich, Canton of Zurich
  - Ospedale Regional Bellinzona e /ID# 151232, Bellinzona
- Turkey (Türkiye) (5):
  - Ankara Univ Medical Faculty /ID# 147443, Ankara
  - Istanbul University Istanbul Medical Faculty /ID# 156040, Istanbul
  - Vehbi Koc vakfi Amerikan Hasta /ID# 147325, Istanbul
  - Dokuz Eylul University /ID# 147442, Izmir
  - Ondokuz mayis University Facul /ID# 147326, Samsun
- United Kingdom (4):
  - Blackpool Teaching Hosp NHS /ID# 149581, Blackpool
  - Univ Hosp Bristol NHS Foundati /ID# 147647, Bristol
  - Southampton General Hospital /ID# 147646, Southampton
  - The Royal Wolverhampton NHS Tr /ID# 147945, Wolverhampton

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing, please refer to the link below.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information on the process, or to submit a request, visit the following link.
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- [Derived] Kater AP, Arslan O, Demirkan F, Herishanu Y, Ferhanoglu B, Diaz MG, Leber B, Montillo M, Panayiotidis P, Rossi D, Skarbnik A, Tempescul A, Turgut M, Mellink CH, van der Kevie-Kersemaekers AF, Lanham S, Sale B, Del Rio L, Popovic R, Chyla BJ, Busman T, Komlosi V, Wang X, Sail K, Pena GE, Vizkelety T, Forconi F. Activity of venetoclax in patients with relapsed or refractory chronic lymphocytic leukaemia: analysis of the VENICE-1 multicentre, open-label, single-arm, phase 3b trial. Lancet Oncol. 2024 Apr;25(4):463-473. doi: 10.1016/S1470-2045(24)00070-6. Epub 2024 Mar 8. PMID 38467131

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 59 sites in 19 countries. The primary analysis of results occurred after all participants completed the Week 48 disease assessment, with a data cut-off date of 30 June 2019.
Groups:
- Venetoclax: Participants received venetoclax on a once daily (QD) dosing schedule for up to 108 weeks. The starting dose was 20 mg daily, increasing over a period of 5 weeks up to the daily dose of 400 mg.
  In countries where venetoclax was not commercially available, participants who continued to derive benefit after 2 years of treatment could extend their treatment for up to two additional years plus one additional year until the venetoclax extension study was open.
Period: Overall Study
Arm/Group | Venetoclax
Started | 258
Completed (Completed survival follow up period or beyond 108 weeks of treatment) | 124
Not Completed | 134
Not completed — Death | 70
Not completed — Withdrawal by Subject | 2
Not completed — Lost to Follow-up | 3
Not completed — Transitioned to Long-term Extension Study M19-388 (NCT03844048) | 49
Not completed — Other | 10

BASELINE CHARACTERISTICS:
Groups:
- Venetoclax: Participants received venetoclax on a once daily dosing schedule for up to 108 weeks. The starting dose was 20 mg daily, increasing over a period of 5 weeks up to the daily dose of 400 mg. Participants who continued to derive benefit after 2 years of treatment may have continued venetoclax therapy for up to 3 additional years.
Arm/Group | Venetoclax
Number analyzed (Participants) | 258
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.7 (9.04)
Age, Customized [Count of Participants; unit: Participants]
  < 65 years | 94
  >= 65 years | 164
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78
  Male | 180
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9
  Not Hispanic or Latino | 248
  Unknown or Not Reported | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 252
  Black or African American | 3
  Asian | 2
  Missing | 1
Geographic Region [Count of Participants; unit: Participants]
  Europe | 161
  North America | 28
  Rest of the World | 69
Prior Treatment With B-cell Receptor Inhibitor (BCRi) [Count of Participants; unit: Participants]
  BCRi-naive | 191
  BCRi-exposed | 67

OUTCOME MEASURES:

1. Primary Outcome: Complete Remission Rate in Participants Not Previously Treated With BCRi Therapy - Primary Analysis
Description: Complete remission rate is defined as the percentage of participants achieving a best response of complete remission (CR) or complete remission with incomplete marrow recovery (CRi) assessed by the investigator based on 2008 Modified International Workshop for Chronic Lymphocytic Leukemia National Cancer Institute-Working Group (IWCLL NCI-WG) criteria.
  CR required all of the following:
  * Peripheral blood lymphocytes < 4000/μL
  * Absence of lymphadenopathy by physical examination and computed tomography scan
  * No hepatomegaly or splenomegaly by physical examination
  * Absence of disease or constitutional symptoms (unexplained fevers > 38°C, drenching night sweats, > 10% weight loss in last 6 months)
  * Blood counts above the following:
    * Neutrophils > 1500/μL
    * Platelets > 100,000/μL
    * Hemoglobin > 110 g/L
  * Bone marrow at least normocellular for age, < 30% lymphocytes.
  CRi was defined as for CR but with persistent cytopenia apparently unrelated to CLL but related to drug toxicity.
Time Frame: From first dose of study drug until the last participant completed Week 48 assessments (data cut-off date 30 June 2019); overall median time on follow-up was 23.2 months.
Population: All enrolled participants treated with at least one dose of venetoclax who had not previously received treatment with BCRi
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Venetoclax
Number analyzed (Participants) | 191
percentage of participants | 35.1 [28.3 to 42.3]
Statistical Analysis 1: Comparison: Venetoclax; The null hypothesis stated that the CR rate for BCRi-naïve participants would be ≤ 6%, based on the CR rate reported for current therapies at the time the study was designed, with an alternative hypothesis that the CR rate would be > 6%. If the p-value for this test was < 0.025, the null hypothesis would be rejected; Test type: Superiority; p < 0.001, Binomial test

2. Secondary Outcome: Complete Remission Rate in Participants Previously Treated With BCRi Therapy - Primary Analysis
Description: Complete remission rate is defined as the percentage of participants achieving a best response of complete remission (CR) or complete remission with incomplete marrow recovery (CRi) assessed by the investigator based on 2008 modified IWCLL NCI-WG criteria.
  CR required all of the following:
  * Peripheral blood lymphocytes < 4000/μL
  * Absence of lymphadenopathy by physical examination and computed tomography scan
  * No hepatomegaly or splenomegaly by physical examination
  * Absence of disease or constitutional symptoms (unexplained fevers > 38°C, drenching night sweats, > 10% weight loss in last 6 months)
  * Blood counts above the following:
    * Neutrophils > 1500/μL
    * Platelets > 100,000/μL
    * Hemoglobin > 110 g/L
  * Bone marrow at least normocellular for age, < 30% lymphocytes
  CRi was defined as for CR but with persistent cytopenia apparently unrelated to CLL but related to drug toxicity.
Time Frame: as for outcome 1
Population: All enrolled participants treated with at least one dose of venetoclax who were previously treated with BCRi
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Venetoclax
Number analyzed (Participants) | 67
percentage of participants | 25.4 [15.5 to 37.5]

3. Secondary Outcome: Overall Response Rate (ORR) - Primary Analysis
Description: Overall response rate was defined as the percentage of participants with an overall best response of CR, CRi, nodular partial remission (nPR), or confirmed partial remission (PR) based on the 2008 modified IWCLL NCI-WG criteria assessed by the investigator.
  CR and CRi are defined above. nPR is defined as for CR but bone marrow nodules could be identified histologically.
  For PR at least 2 of the following must be met:
  * 50% decrease in peripheral blood lymphocyte count from the Baseline value;
  * 50% reduction in lymphadenopathy;
  * 50% reduction in the size of the liver and/or spleen (if abnormal prior to therapy);
  In addition at least 1 of the following criteria must be met:
  * Neutrophils > 1,500/μL or ≥ 50% improvement over Baseline;
  * Platelets > 100,000/μL or ≥ 50% improvement over Baseline;
  * Hemoglobin > 11.0 g/dL or ≥ 50% improvement over Baseline without transfusions or exogenous growth factors.
  PR must have been confirmed at least 7 weeks later.
Time Frame: as for outcome 1
Population: All enrolled participants treated with at least one dose of venetoclax
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Venetoclax
Number analyzed (Participants) | 258
percentage of participants | 79.8 [74.4 to 84.6]

4. Secondary Outcome: Duration of Overall Response (DOR) - Primary Analysis
Description: Duration of response was defined as the time from the date of first response (CR, CRi, nPR, or PR) to the earliest date that progressive disease (PD) was objectively documented (radiographic or clinical) or death. Duration of response was analyzed by Kaplan-Meier (K-M) methodology. If a participant was still responding the data were censored at the date of the last available disease assessment prior to the data cutoff date.
Time Frame: as for outcome 1
Population: Enrolled participants treated with at least one dose of venetoclax who had an overall response of CR, CRi, nPR, or confirmed PR.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Venetoclax
Number analyzed (Participants) | 205
months | 25.2 [23.0 to 25.2]

5. Secondary Outcome: Time to Progression (TTP) - Primary Analysis
Description: Time to progression was defined as the time from the date of first dose of venetoclax to the date of earliest PD (radiographic or clinical). Participants who did not experience disease progression were censored at the date of the last available disease assessment prior to the data cutoff date; participants with no post-baseline disease assessments were censored at the first dose date plus 1 day. Time to progression was estimated using Kaplan-Meier methodology.
Time Frame: as for outcome 1
Population: Enrolled participants treated with at least one dose of venetoclax
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Venetoclax
Number analyzed (Participants) | 258
months | 30.5 [29.6 to 30.5]

6. Secondary Outcome: Progression-Free Survival (PFS) - Primary Analysis
Description: Progression-free survival (PFS) was defined as the time from the date of first dose of venetoclax to the date of earliest PD (radiographic or clinical) or death. Participants who did not experience disease progression or death were censored at the date of the last available disease assessment prior to the data cutoff date; participants with no post-baseline tumor assessment or clinical assessment for progression were censored at the date of first dose plus 1 day. Progression-free survival was analyzed by Kaplan-Meier methodology.
Time Frame: as for outcome 1
Population: Enrolled participants treated with at least one dose of venetoclax
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Venetoclax
Number analyzed (Participants) | 258
months | 30.5 [28.6 to 30.5]

7. Secondary Outcome: Overall Survival (OS) - Primary Analysis
Description: Overall survival (time to death) was defined as the time from the first dose date of venetoclax to the date of death. If a participant had not died the data were censored at the date when they were last known to be alive prior to the cutoff date. Overall survival was analyzed using Kaplan-Meier methodology.
Time Frame: as for outcome 1
Population: Enrolled participants treated with at least one dose of venetoclax
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Venetoclax
Number analyzed (Participants) | 258
months | NA [NA to NA] — Could not be estimated due to the low number of events

8. Secondary Outcome: Change From Baseline in Functional Assessment of Cancer Therapy - Leukemia Questionnaire (FACT-Leu)
Description: The FACT-Leu is a 44-item, leukemia-specific questionnaire designed to assess health-related quality of life (HRQoL) and leukemia-specific symptoms using a core set of questions (Functional Assessment of Cancer Therapy-General; FACT-G), and a cancer site-specific leukemia subscale. Questions are scored on a scale from 0 (not at all) to 4 (very much).
  FACT-G consists of 27 general items divided into 4 primary HRQoL domains: Physical Well-being (PWB; 7 items; score range 0-28), Social/Family Well-being (SWB; 7 items; score range 0-28), Emotional Well-being (EWB; 6 items; score range 0-24), Functional Well-being (FWB; 7 items; score range 0-28). The leukemia subscale consists of 17 items (score range 0-68) that assess patient concerns relating to leukemia. Three summary scales were calculated: FACT-Trial Outcome Index composed of the PWB, FWB, and leukemia subscale (score range 0-124); FACT-G (score range 0-108) and the FACT-Leu Total (range 0-176). Higher scores reflect better HRQoL.
Time Frame: Baseline and Weeks 48 and 108
Population: All enrolled participants treated with at least one dose of venetoclax with available data at each time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Venetoclax
Number analyzed (Participants) | 205
score on a scale
  Physical well-being - Week 48 | 1.2 (4.07)
  Physical well-being - Week 108: number analyzed (Participants) | 153
  Physical well-being - Week 108 | 0.9 (4.20)
  Social/family well-being - Week 48: number analyzed (Participants) | 203
  Social/family well-being - Week 48 | 0.2 (5.14)
  Social/family well-being - Week 108: number analyzed (Participants) | 151
  Social/family well-being - Week 108 | -0.4 (4.86)
  Emotional well-being - Week 48: number analyzed (Participants) | 202
  Emotional well-being - Week 48 | 2.1 (3.52)
  Emotional well-being - Week 108: number analyzed (Participants) | 154
  Emotional well-being - Week 108 | 1.7 (3.94)
  Functional well-being - Week 48: number analyzed (Participants) | 202
  Functional well-being - Week 48 | 1.8 (5.63)
  Functional well-being - Week 108: number analyzed (Participants) | 153
  Functional well-being - Week 108 | 1.4 (5.67)
  Leukemia subscale - Week 48: number analyzed (Participants) | 202
  Leukemia subscale - Week 48 | 6.8 (7.99)
  Leukemia subscale - Week 108: number analyzed (Participants) | 153
  Leukemia subscale - Week 108 | 6.0 (9.08)
  FACT-G total score - Week 48: number analyzed (Participants) | 200
  FACT-G total score - Week 48 | 5.5 (12.34)
  FACT-G total score - Week 108: number analyzed (Participants) | 148
  FACT-G total score - Week 108 | 3.6 (13.56)
  FACT-leukemia trial outcome index - Week 48: number analyzed (Participants) | 201
  FACT-leukemia trial outcome index - Week 48 | 9.8 (14.23)
  FACT-leukemia trial outcome index - Week 108: number analyzed (Participants) | 150
  FACT-leukemia trial outcome index - Week 108 | 8.2 (15.61)
  FACT-leukemia total score - Week 48: number analyzed (Participants) | 199
  FACT-leukemia total score - Week 48 | 12.3 (18.18)
  FACT-leukemia total score - Week 108: number analyzed (Participants) | 147
  FACT-leukemia total score - Week 108 | 9.5 (20.62)

9. Secondary Outcome: Change From Baseline in Functional Assessment of Chronic Illness Therapy - Fatigue Scale (FACIT-Fatigue)
Description: The FACIT-Fatigue questionnaire measures fatigue and its effect on functioning and daily activities. The FACIT-Fatigue includes 13 items answered on a 5-point rating scale based on a 7-day recall period. Scores range from 0 to 52, with lower scores reflecting greater fatigue.
Time Frame: Baseline and Weeks 48 and 108
Population: All enrolled participants treated with at least one dose of venetoclax with available data at each time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Venetoclax
Number analyzed (Participants) | 205
score on a scale
  Week 48 | 4.9 (9.43)
  Week 108: number analyzed (Participants) | 154
  Week 108 | 3.3 (9.96)

10. Secondary Outcome: Change From Baseline in EuroQoL 5 Dimension 5 Level Questionnaire (EQ-5D-5L) Health Index Score
Description: The EQ-5D-5L is a generic measure of health status consisting of two parts: a descriptive system consisting of 5 items and a visual analog scale (VAS).
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The participant is asked to rate each dimension on 5 levels of severity (1: no problems, 2: slight problems, 3: moderate problems, 4: severe problems, 5: extreme problems).
  The scores for the 5 dimensions are used to compute a single health utility index score representing the general health status of the individual. The health index score ranges from zero (defined as a health state equivalent to being dead) to 1 (full health).
Time Frame: Baseline and Weeks 48 and 108
Population: All enrolled participants treated with at least one dose of venetoclax with available data at each time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Venetoclax
Number analyzed (Participants) | 204
score on a scale
  Week 48 | 0.0 (0.14)
  Week 108: number analyzed (Participants) | 152
  Week 108 | 0.0 (0.15)

11. Secondary Outcome: Change From Baseline in EuroQoL 5 Dimension 5 Level Questionnaire (EQ-5D-5L) Visual Analog Scale Score
Description: The EQ-5D-5L is a generic measure of health status consisting of two parts, a descriptive system consisting of 5 items and a visual analog scale (VAS).
  The VAS assesses the participant's self-rated overall health on a scale from 0 (worst health imaginable) to 100 (best health imaginable).
Time Frame: Baseline and Weeks 48 and 108
Population: All enrolled participants treated with at least one dose of venetoclax with available data at each time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Venetoclax
Number analyzed (Participants) | 204
score on a scale
  Week 48 | 8.5 (14.43)
  Week 108: number analyzed (Participants) | 156
  Week 108 | 7.1 (14.61)

12. Other Pre Specified Outcome: Complete Remission Rate in Participants Not Previously Treated With BCRi Therapy - Final Analysis
Description: Complete remission rate is defined as the percentage of participants achieving a best response of complete remission (CR) or complete remission with incomplete marrow recovery (CRi) assessed by the investigator based on 2008 modified IWCLL NCI-WG criteria.
  CR required all of the following:
  * Peripheral blood lymphocytes < 4000/μL
  * Absence of lymphadenopathy by physical examination and computed tomography scan
  * No hepatomegaly or splenomegaly by physical examination
  * Absence of disease or constitutional symptoms (unexplained fevers > 38°C, drenching night sweats, > 10% weight loss in last 6 months)
  * Blood counts above the following:
    * Neutrophils > 1500/μL
    * Platelets > 100,000/μL
    * Hemoglobin > 110 g/L
  * Bone marrow at least normocellular for age, < 30% lymphocytes.
  CRi was defined as for CR but with persistent cytopenia apparently unrelated to CLL but related to drug toxicity.
Time Frame: From first dose of study drug until the end of study; overall median time on follow-up was 49.5 months.
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Venetoclax
Number analyzed (Participants) | 191
percentage of participants | 34.6 [27.8 to 41.8]
Statistical Analysis 1: Comparison: Venetoclax; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, Binomial test

13. Other Pre Specified Outcome: Complete Remission Rate in Participants Previously Treated With BCRi Therapy - Final Analysis
Description: as for outcome 2
Time Frame: From first dose of study drug until the end of study; overall median time on follow-up was 49.5 months.
Population: All enrolled participants treated with at least one dose of venetoclax who were previously treated with BCRi
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Venetoclax
Number analyzed (Participants) | 67
percentage of participants | 26.9 [16.8 to 39.1]

14. Other Pre Specified Outcome: Overall Response Rate (ORR) - Final Analysis
Description: as for outcome 3
Time Frame: From first dose of study drug until the end of study; overall median time on follow-up was 49.5 months.
Population: All enrolled participants treated with at least one dose of venetoclax
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Venetoclax
Number analyzed (Participants) | 258
percentage of participants | 79.8 [74.4 to 84.6]

15. Other Pre Specified Outcome: Duration of Overall Response (DOR) - Final Analysis
Description: as for outcome 4
Time Frame: From first dose of study drug until the end of study; overall median time on follow-up was 49.5 months.
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Venetoclax
Number analyzed (Participants) | 205
months | 25.1 [19.4 to 28.6]

16. Other Pre Specified Outcome: Time to Progression (TTP) - Final Analysis
Description: as for outcome 5
Time Frame: From first dose of study drug until the end of study; overall median time on follow-up was 49.5 months.
Population: Enrolled participants treated with at least one dose of venetoclax
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Venetoclax
Number analyzed (Participants) | 258
months | 28.3 [23.4 to 32.6]

17. Other Pre Specified Outcome: Progression-Free Survival (PFS) - Final Analysis
Description: as for outcome 6
Time Frame: From first dose of study drug until the end of study; overall median time on follow-up was 49.5 months.
Population: Enrolled participants treated with at least one dose of venetoclax
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Venetoclax
Number analyzed (Participants) | 258
months | 28.3 [22.2 to 30.5]

18. Other Pre Specified Outcome: Overall Survival (OS) - Final Analysis
Description: as for outcome 7
Time Frame: From first dose of study drug until the end of study; overall median time on follow-up was 49.5 months.
Population: Enrolled participants treated with at least one dose of venetoclax
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Venetoclax
Number analyzed (Participants) | 258
months | NA [NA to NA] — Could not be estimated due to the low number of events

19. Other Pre Specified Outcome: Minimal Residual Disease (MRD) Negativity Rate - Primary Analysis
Description: The MRD negativity rate is defined as the percentage of participants who had MRD negative status with less than one CLL cell per 10,000 leukocytes (< 10-⁴) in peripheral blood and bone marrow. MRD was evaluated using next-generation sequencing. Per protocol, peripheral blood MRD assessments were to be collected from all participants at Week 24 and Week 48 and at the time the bone marrow assessment for confirmation of CR/CRi, and bone marrow (BM) MRD assessments were to be collected for participants undergoing a bone marrow procedure for confirmation of CR/CRi. Participants with no blood or BM MRD assessments were included in the calculation of MRD negativity rate as not having MRD negative status.
Time Frame: as for outcome 1
Population: All enrolled participants who received at least one dose of venetoclax
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Venetoclax
Number analyzed (Participants) | 258
percentage of participants
  Peripheral blood | 39.9 [33.9 to 46.2]
  Bone marrow | 9.7 [6.4 to 14.0]

20. Other Pre Specified Outcome: Minimal Residual Disease (MRD) Negativity Rate - Final Analysis
Description: as for outcome 19
Time Frame: From first dose of study drug until the end of study; overall median time on follow-up was 49.5 months.
Population: All enrolled participants who received at least one dose of venetoclax
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Venetoclax
Number analyzed (Participants) | 258
percentage of participants
  Peripheral blood | 40.3 [34.3 to 46.6]
  Bone marrow | 10.5 [7.0 to 14.9]

ADVERSE EVENTS:
Time Frame: All-cause mortality are reported up to the end of the study; median time on study was 210 weeks. Adverse events are reported from the first dose of venetoclax up to 30 days after the last dose of venetoclax; Median (minimum, maximum) duration of treatment was 108 (0.1, 254.6) weeks.
Arm/Group | Venetoclax
All-Cause Mortality (participants affected / at risk) | 70/258
Serious Adverse Events (participants affected / at risk) | 136/258
Other Adverse Events (participants affected / at risk) | 246/258
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Venetoclax (N=258)
ANAEMIA (Blood and lymphatic system disorders) | 5 (5)
APLASIA PURE RED CELL (Blood and lymphatic system disorders) | 1 (1)
AUTOIMMUNE HAEMOLYTIC ANAEMIA (Blood and lymphatic system disorders) | 3 (6)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 15 (18)
GRANULOMATOUS LYMPHADENITIS (Blood and lymphatic system disorders) | 1 (1)
HAEMOLYSIS (Blood and lymphatic system disorders) | 1 (1)
INTRAVASCULAR HAEMOLYSIS (Blood and lymphatic system disorders) | 1 (2)
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 1 (1)
NEUTROPENIA (Blood and lymphatic system disorders) | 4 (4)
PANCYTOPENIA (Blood and lymphatic system disorders) | 2 (2)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 3 (4)
AORTIC VALVE STENOSIS (Cardiac disorders) | 1 (1)
ATRIAL FIBRILLATION (Cardiac disorders) | 1 (1)
ATRIOVENTRICULAR BLOCK (Cardiac disorders) | 1 (1)
BIFASCICULAR BLOCK (Cardiac disorders) | 1 (1)
BRADYCARDIA (Cardiac disorders) | 1 (1)
CARDIAC ARREST (Cardiac disorders) | 1 (1)
CARDIAC FAILURE (Cardiac disorders) | 2 (2)
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 2 (2)
CORONARY ARTERY DISEASE (Cardiac disorders) | 2 (2)
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1)
HYDROCELE (Congenital, familial and genetic disorders) | 1 (1)
DEAFNESS NEUROSENSORY (Ear and labyrinth disorders) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 3 (3)
ASCITES (Gastrointestinal disorders) | 1 (1)
DIARRHOEA (Gastrointestinal disorders) | 5 (5)
DIVERTICULUM INTESTINAL HAEMORRHAGIC (Gastrointestinal disorders) | 1 (1)
INGUINAL HERNIA (Gastrointestinal disorders) | 2 (2)
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 (1)
RECTAL PERFORATION (Gastrointestinal disorders) | 1 (1)
VOMITING (Gastrointestinal disorders) | 1 (1)
CHEST PAIN (General disorders) | 1 (1)
FATIGUE (General disorders) | 1 (1)
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 1 (1)
MALAISE (General disorders) | 2 (2)
MUCOSAL HAEMORRHAGE (General disorders) | 1 (1)
MULTIPLE ORGAN DYSFUNCTION SYNDROME (General disorders) | 2 (3)
PYREXIA (General disorders) | 11 (12)
BILE DUCT STONE (Hepatobiliary disorders) | 1 (1)
BILIARY COLIC (Hepatobiliary disorders) | 1 (1)
CHOLANGITIS (Hepatobiliary disorders) | 1 (1)
CHOLELITHIASIS (Hepatobiliary disorders) | 1 (1)
GALLBLADDER NECROSIS (Hepatobiliary disorders) | 1 (1)
HEPATIC CIRRHOSIS (Hepatobiliary disorders) | 1 (1)
DRUG HYPERSENSITIVITY (Immune system disorders) | 1 (1)
HYPERSENSITIVITY (Immune system disorders) | 1 (1)
ABSCESS LIMB (Infections and infestations) | 1 (1)
ARTHRITIS BACTERIAL (Infections and infestations) | 1 (1)
BRONCHIOLITIS (Infections and infestations) | 1 (1)
BRONCHITIS (Infections and infestations) | 2 (2)
CELLULITIS (Infections and infestations) | 2 (2)
COVID-19 (Infections and infestations) | 2 (3)
DIVERTICULITIS (Infections and infestations) | 1 (1)
ENDOPHTHALMITIS (Infections and infestations) | 1 (1)
EPIDIDYMITIS (Infections and infestations) | 1 (1)
ESCHERICHIA INFECTION (Infections and infestations) | 1 (2)
GASTROENTERITIS (Infections and infestations) | 2 (2)
HERPES ZOSTER (Infections and infestations) | 2 (2)
INFLUENZA (Infections and infestations) | 3 (3)
LOCALISED INFECTION (Infections and infestations) | 1 (1)
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 4 (4)
NEUTROPENIC SEPSIS (Infections and infestations) | 1 (1)
OSTEOMYELITIS (Infections and infestations) | 1 (1)
PNEUMONIA (Infections and infestations) | 21 (30)
PNEUMONIA BACTERIAL (Infections and infestations) | 1 (1)
PROGRESSIVE MULTIFOCAL LEUKOENCEPHALOPATHY (Infections and infestations) | 1 (1)
PYELONEPHRITIS (Infections and infestations) | 1 (1)
RESPIRATORY SYNCYTIAL VIRUS INFECTION (Infections and infestations) | 2 (2)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 (2)
SEPSIS (Infections and infestations) | 1 (1)
SEPTIC SHOCK (Infections and infestations) | 2 (2)
SKIN INFECTION (Infections and infestations) | 1 (1)
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 1 (1)
TONSILLITIS BACTERIAL (Infections and infestations) | 1 (1)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 (2)
UROSEPSIS (Infections and infestations) | 1 (1)
CLAVICLE FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
CONTUSION (Injury, poisoning and procedural complications) | 1 (1)
FALL (Injury, poisoning and procedural complications) | 2 (4)
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
HEAD INJURY (Injury, poisoning and procedural complications) | 1 (1)
HIP FRACTURE (Injury, poisoning and procedural complications) | 2 (2)
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
INFUSION RELATED REACTION (Injury, poisoning and procedural complications) | 1 (1)
PELVIC FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 3 (3)
BLOOD BILIRUBIN INCREASED (Investigations) | 1 (1)
BLOOD CREATININE INCREASED (Investigations) | 2 (2)
BLOOD LACTATE DEHYDROGENASE INCREASED (Investigations) | 4 (4)
BLOOD PHOSPHORUS INCREASED (Investigations) | 1 (1)
BLOOD POTASSIUM INCREASED (Investigations) | 3 (3)
GENERAL PHYSICAL CONDITION ABNORMAL (Investigations) | 1 (1)
PLATELET COUNT DECREASED (Investigations) | 1 (1)
WEIGHT DECREASED (Investigations) | 2 (2)
CACHEXIA (Metabolism and nutrition disorders) | 1 (1)
DIABETES MELLITUS (Metabolism and nutrition disorders) | 1 (1)
FLUID RETENTION (Metabolism and nutrition disorders) | 1 (1)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPERKALAEMIA (Metabolism and nutrition disorders) | 4 (7)
HYPERPHOSPHATAEMIA (Metabolism and nutrition disorders) | 3 (4)
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 1 (1)
TUMOUR LYSIS SYNDROME (Metabolism and nutrition disorders) | 2 (2)
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
HAEMATOMA MUSCLE (Musculoskeletal and connective tissue disorders) | 1 (1)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (2)
OSTEOPOROSIS (Musculoskeletal and connective tissue disorders) | 1 (1)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 (1)
SPINAL PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
ADENOMA BENIGN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
ADRENAL ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
BLADDER CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
CENTRAL NERVOUS SYSTEM LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
CHRONIC LYMPHOCYTIC LEUKAEMIA TRANSFORMATION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2)
DIFFUSE LARGE B-CELL LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
INFECTED NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
LUNG ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
MYELODYSPLASTIC SYNDROME (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4)
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
RECTAL ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
SKIN NEOPLASM BLEEDING (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
SQUAMOUS CELL CARCINOMA OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
ATAXIA (Nervous system disorders) | 1 (1)
DIZZINESS (Nervous system disorders) | 1 (1)
DYSARTHRIA (Nervous system disorders) | 1 (1)
FACIAL PARALYSIS (Nervous system disorders) | 1 (1)
HAEMORRHAGE INTRACRANIAL (Nervous system disorders) | 1 (1)
ISCHAEMIC STROKE (Nervous system disorders) | 2 (3)
METABOLIC ENCEPHALOPATHY (Nervous system disorders) | 1 (1)
SCIATICA (Nervous system disorders) | 1 (1)
SEIZURE (Nervous system disorders) | 1 (1)
SOMNOLENCE (Nervous system disorders) | 1 (1)
SUBARACHNOID HAEMORRHAGE (Nervous system disorders) | 1 (1)
SYNCOPE (Nervous system disorders) | 2 (3)
CONFUSIONAL STATE (Psychiatric disorders) | 2 (3)
DEPRESSION (Psychiatric disorders) | 1 (1)
MENTAL STATUS CHANGES (Psychiatric disorders) | 1 (2)
READING DISORDER (Psychiatric disorders) | 1 (1)
BLADDER MASS (Renal and urinary disorders) | 1 (1)
BENIGN PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 3 (3)
PROSTATIC PAIN (Reproductive system and breast disorders) | 1 (1)
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 2 (2)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 1 (1)
ATELECTASIS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
BRONCHIECTASIS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 (2)
COUGH (Respiratory, thoracic and mediastinal disorders) | 3 (3)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 5 (5)
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 1 (1)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
LUNG DISORDER (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PHARYNGEAL DISORDER (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PHARYNGEAL SWELLING (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 3 (4)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 2 (2)
PULMONARY HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 1 (2)
PARANEOPLASTIC PEMPHIGUS (Skin and subcutaneous tissue disorders) | 1 (1)
RASH (Skin and subcutaneous tissue disorders) | 1 (1)
SKIN ULCER (Skin and subcutaneous tissue disorders) | 2 (2)
ANEURYSM (Vascular disorders) | 1 (1)
AORTIC INTRAMURAL HAEMATOMA (Vascular disorders) | 1 (1)
DEEP VEIN THROMBOSIS (Vascular disorders) | 1 (1)
HYPERTENSIVE CRISIS (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Venetoclax (N=258)
ANAEMIA (Blood and lymphatic system disorders) | 57 (84)
NEUTROPENIA (Blood and lymphatic system disorders) | 108 (251)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 53 (88)
ABDOMINAL PAIN (Gastrointestinal disorders) | 21 (23)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 13 (17)
CONSTIPATION (Gastrointestinal disorders) | 34 (42)
DIARRHOEA (Gastrointestinal disorders) | 95 (170)
DYSPEPSIA (Gastrointestinal disorders) | 13 (13)
NAUSEA (Gastrointestinal disorders) | 69 (98)
VOMITING (Gastrointestinal disorders) | 20 (24)
ASTHENIA (General disorders) | 32 (41)
FATIGUE (General disorders) | 45 (56)
OEDEMA PERIPHERAL (General disorders) | 13 (17)
PYREXIA (General disorders) | 43 (56)
HERPES ZOSTER (Infections and infestations) | 14 (17)
INFLUENZA (Infections and infestations) | 14 (14)
NASOPHARYNGITIS (Infections and infestations) | 39 (62)
PNEUMONIA (Infections and infestations) | 16 (19)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 47 (68)
URINARY TRACT INFECTION (Infections and infestations) | 25 (39)
FALL (Injury, poisoning and procedural complications) | 13 (14)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 13 (15)
NEUTROPHIL COUNT DECREASED (Investigations) | 28 (47)
PLATELET COUNT DECREASED (Investigations) | 21 (27)
WEIGHT DECREASED (Investigations) | 22 (25)
DECREASED APPETITE (Metabolism and nutrition disorders) | 24 (29)
HYPERKALAEMIA (Metabolism and nutrition disorders) | 21 (31)
HYPERPHOSPHATAEMIA (Metabolism and nutrition disorders) | 20 (23)
HYPERURICAEMIA (Metabolism and nutrition disorders) | 17 (17)
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 15 (19)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 15 (20)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 37 (50)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 34 (36)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 17 (20)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 14 (17)
DIZZINESS (Nervous system disorders) | 20 (26)
HEADACHE (Nervous system disorders) | 27 (29)
INSOMNIA (Psychiatric disorders) | 25 (27)
COUGH (Respiratory, thoracic and mediastinal disorders) | 52 (63)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 23 (26)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 14 (15)
DRY SKIN (Skin and subcutaneous tissue disorders) | 17 (22)
PRURITUS (Skin and subcutaneous tissue disorders) | 25 (29)
RASH (Skin and subcutaneous tissue disorders) | 20 (33)
HYPERTENSION (Vascular disorders) | 29 (34)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2020-10-12): https://cdn.clinicaltrials.gov/large-docs/11/NCT02756611/Prot_002.pdf
  • Statistical Analysis Plan (2018-12-20): https://cdn.clinicaltrials.gov/large-docs/11/NCT02756611/SAP_000.pdf